CLINICAL TRIAL: NCT05970874
Title: Musculoskeletal Pain in Pregnant Infected With COVID-19, Evaluation of Fatigue and Muscle Grip Strength
Brief Title: Evaluation of Hand Grip Strength in Pregnant COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 06-2022/10
Record Dates: First submitted 2023-07-30; First posted 2023-08-01 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: COVID-19; Pregnancy Related
Keywords: COVID-19; Musculoskeletal Symptom; Hand Grip Muscle Streng
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pregnant covid 19 patients: pregnant covid 19 patients
  Interventions: Device: Hand grip strength measureme

INTERVENTIONS:
Device: Hand grip strength measureme — Hand grip strength (HSG) was measured in kg with the CAMRY Digital Hand Dynamometer (Model No. EH101, CAMRY).

SUMMARY:
It was presented as a cross-sectional, single-center, retrospective case series. Pregnant women with a positive Polymerase Chain Reaction (PCR) diagnosis of Covid 19 were included in the study. The relationship between patients' musculoskeletal symptoms and signs and hand grip strength was investigated.

DETAILED DESCRIPTION:
Covid 19 is the disease defined for strains infected with severe acute respiratory syndrome coronavirus 2(Sars-CoV-2). Hand grip strength is a non-invasive, easily applicable, objective parameter. It was presented as a cross-sectional, single-center, retrospective case series. Pregnant women with a positive Polymerase Chain Reaction (PCR) diagnosis of Covid 19 were included in the study. The relationship between patients' musculoskeletal symptoms and signs and hand grip strength was investigated.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with a positive Polymerase Chain Reaction (PCR) diagnosis of Covid 19

Exclusion Criteria:

* Those with orthopedic defects in the dominant hand and wrist and those with hand, wrist and shoulder involvement on the side of the measurement related to rheumatological diseases were excluded from the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: pregnant covid 19 patients
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Hand grip strength assessment | The first 24 hours after admission to the service.
  Hand grip strength assessment in pregnancy Covid 19.

SECONDARY OUTCOMES:
symptoms | The first 24 hours after admission to the service.
  Common symptoms of pregnant Covid 19 patients.
laboratory findings | The first 24 hours after admission to the service.
  Common laboratory findings of pregnant Covid 19 patients.
Vaccine | pre-infection period was questioned
  Vaccine rate of pregnant Covid 19 patients.
Smoking | pre-infection period was questioned
  Smoking rate of pregnant Covid 19 patients.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Toprak, Principal Investigator — dr.tprk@hotmail.com
Locations (1):
- Hatice Toprak, Karaman, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No